CLINICAL TRIAL: NCT04566276
Title: A Phase 1/2, Dose-finding Study to Evaluate Safety, Tolerability, and Immunogenicity of the ChulaCov19 Vaccine in Healthy Adults
Brief Title: ChulaCov19 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Chula Vaccine Research Center (ChulaVRC), Bangkok, Thailand (Unknown); Center of Excellence in Vaccine Research and Development, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand (Unknown); Chula Clinical Research Center (Chula CRC), King Chulalongkorn Memorial Hospital, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand (Unknown); King Chulalongkorn Memorial Hospital (KCMH), Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand (Unknown); Mahidol University (Other); National Vaccine Institute, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: ChulaVac 001
Record Dates: First submitted 2020-09-15; First posted 2020-09-28 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Vaccine; Safety Issues
Keywords: tolerability; reactivity; immunogenicity; healthy adults; healthy elderlies; coronavirus disease 2019; SARS-CoV-2-specific serum neutralising antibody titer; SARS-CoV-2-surrogate viral neutralising antibody; SARS-Cov2 spike protein-binding IgG antibody titer; SARS-Cov2 spike protein-specific CD4+ and CD8+ T-cells responses; IFNγ enzyme-linked immune absorbent spot (ELISpot); SARS-Cov2 spike protein-specific Th1/Th2 polarisation; novel lipid nanoparticles (LNPs)-encapsulated mRNA-based vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChulaCov19 vaccine

STUDY DESIGN:
Intervention Model Description: Phase 1: Group 1 (healthy adults aged 18 to 55 years) and Group 2 (elderlies aged 56 to 75 years) will be enrolled sequentially in an ascending dose fashion (10 µg, 25 µg, 50 µg). Up to 36 eligible healthy volunteers for each of the 2 age groups will be enrolled into 1 of 3 treatment cohorts (12 participants/ cohort). For each cohort, if only 1 participant withdraws prior to the second vaccination, no replacement is deemed necessary. For each cohort, if more than 1 participant withdraws prior to the second vaccination all withdrawn participants will be replaced.
  Phase 2: The Phase 2 adult cohorts will include adults between 18 and 59 years of age (inclusive). Participants in the Phase 2 will be enrolled into at least 1 dose level cohort with a vaccination dose of 50 ug which was determined by DSMB and SRPT review and approval of the applicable Phase 1 data. Phase 2 treatment group will consist of participants randomly assigned to active treatment versus placebo in a ratio of 4:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Adult Cohort 1: 10 µg (Experimental): 12 healthy adults aged 18-55 years will receive 10 µg of the vaccine IM
  Interventions: Biological: ChulaCov19 vaccine
- Adult Cohort 2: 25 µg (Experimental): 12 healthy adults aged 18-55 years will receive 25 µg of the vaccine IM
  Interventions: Biological: ChulaCov19 vaccine
- Adult Cohort 3: 50 µg (Experimental): 12 healthy adults aged 18-55 years will receive 50 µg of the vaccine IM
  Interventions: Biological: ChulaCov19 vaccine
- Elderly Cohort 1 :10 µg (Experimental): 12 elderlies aged 56-75 years will receive 10 µg of the vaccine IM
  Interventions: Biological: ChulaCov19 vaccine
- Elderly Cohort 2: 25 µg (Experimental): 12 elderlies aged 56-75 years will receive 25 µg of the vaccine IM
  Interventions: Biological: ChulaCov19 vaccine
- Elderly Cohort 3: 50 µg (Experimental): 12 elderlies aged 56-75 years will receive 50 µg of the vaccine IM
  Interventions: Biological: ChulaCov19 vaccine
- Phase 2: ChulaCov19 vaccine Dose 50 ug (Experimental): adults between 18 and 59 years of age will receive 2 IM ChulaCov19 vaccine Dose 50 ug vaccinations; administered 21days apart (on Day 1 and Day 22 ±3)
  Interventions: Biological: ChulaCov19 vaccine
- Phase 2: Placebo (Other): adults between 18 and 59 years of age will receive 2 IM saline vaccinations; administered 21days apart (on Day 1 and Day 22 ±3)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ChulaCov19 vaccine — SARS-Cov2 Wild-type S-spike mRNA/ lipid nanoparticle (LNP) vaccine
  Arms: Adult Cohort 1: 10 µg; Adult Cohort 2: 25 µg; Adult Cohort 3: 50 µg; Elderly Cohort 1 :10 µg; Elderly Cohort 2: 25 µg; Elderly Cohort 3: 50 µg; Phase 2: ChulaCov19 vaccine Dose 50 ug
Other: Placebo — Saline
  Arms: Phase 2: Placebo

SUMMARY:
This study will be conducted in 2 phases. Phase 1 of this study will be a single-centre, open label, dose escalation first in human (FIH) study conducted in 2 groups of healthy participants. Group 1 will enrol adults aged 18-55 years (inclusive); Group 2 will enroll elderly adults (elderly) aged 56-75 years (inclusive).

Phase 2 of this study will be a single centre, the proposed design will be observer-blind, placebo-controlled study to assess the safety, reactogenicity, and immunogenicity of ChulaCov19 vaccine in healthy adults (18-75 years of age inclusive).

DETAILED DESCRIPTION:
This study will be conducted as a combined phase 1/2 study in healthy participants.

The first phase of the study will evaluate the safety, tolerability, and reactogenicity of escalating doses (10 µg, 25 µg, and 50 µg) of the ChulaCov19 vaccine, administered intramuscularly (IM) according to a repeat vaccination schedule (given 21 days apart) in healthy adults aged 18-55 years and in elderly adults aged 56-75 years, up to Visit 10 (Day 50 ±3).

The second phase of the study will evaluate the safety, tolerability, and reactogenicity of escalating doses of the ChulaCov19 vaccine, administered intramuscularly (IM) according to a repeat vaccination schedule (given 21 days apart) in healthy adults aged 18--75 years, up to Visit 10 (Day 50 ±3). The study will also evaluate the immunogenicity measured as neutralising antibody titre (measured by Micro-viral neutralising test [MicroVNT]) following repeat vaccination of escalating doses of the ChulaCov19 vaccine, administered IM according to a repeat vaccination schedule (given 21 days apart) in healthy adults aged 18-75 years, at Visit 9 (Day 29 +3).

ELIGIBILITY:
Participants who meet all the following criteria at Screening are eligible to participate in the study:

Inclusion criteria:

1. Participants must be able to communicate effectively with study personnel and considered reliable, willing, and cooperative in terms of compliance with the protocol requirements.
2. Participants must sign the written informed consent form prior to undertaking any protocol related procedures.
3. Participants must have a body mass index (BMI) at Screening, calculated as the body mass divided (in kilograms [kg]) by the square of the body height (in metres [m]) of 18.0-30.0 kg/m2, inclusive.
4. Participants must have haematology, clinical chemistry, coagulation (for all participants in Phase 1, and, only if applicable, for participants in Phase 2), and urinalysis test results that are not deviating from the normal reference range by age and gender to a clinically relevant extent at Screening.
5. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), practice true abstinence or, if engaged in sexual relations with a female of child-bearing potential, the participants and their partner must use an acceptable, highly effective, double-barrier contraceptive method* from Screening and for a period of at least 60 days after the last dose of investigational vaccine.
6. Women of child-bearing potential must practice true abstinence or, if engaged in sexual relations with a male, they must agree to use highly effective (failure rate of < 1% per year when used consistently and correctly), double-barrier contraceptive measures* throughout the study and intend to continue use of contraception for at least 60 days following the last vaccination.

   * The PI is to assess the adequacy of methods of contraception on a case-by-case basis. These criteria do not apply if the participants are in a same-sex relationship.
7. Women of child-bearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [β-HCG]) at Screening and a negative urine-based test within 24 hours prior to each investigational vaccine administration.
8. Women of non-child-bearing potential must:

   1. be classified as being postmenopausal (defined as having a history of amenorrhea of at least one year), or
   2. where history of amenorrhea is less than one year, female participants must have a follicle stimulating hormone (FSH) level > 40 milli-international units per milliliter (mIU/mL), or
   3. have a documented status of being surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation/salpingectomy).
9. Participants must be in general good health based on medical history and physical examination, as determined by the PI, at Screening.
10. Body temperature must be less than 37.8ºC, at Screening.
11. Pulse must be no greater than 100 beats per minute, at Screening.
12. Systolic blood pressure (SBP) must be between 85 to 150 millimetres of mercury (mm Hg), inclusive, at Screening.
13. Participants must agree to refrain from donating blood, plasma, ovules, sperm, or organs during the whole study.

    Adult Participants (Group 1 of Phase 1) only
14. Must be a male or female aged 18-55 years (inclusive) at the time of enrolment.

    Elderly Participants (Group 2 of Phase 1) only
15. Must be a male or female aged 56-75 years (inclusive) at the time of enrolment.

    Participants for Phase 2 only
16. Must be a male or female aged 18 -59 years (inclusive) at the time of enrolment.

Exclusion Criteria

The presence of any of the following criteria will constitute cause for the exclusion of the participant:

1. Presence of clinically significant medical history, unstable chronic or acute disease, or physical, or laboratory findings that, in the opinion of the PI may potentially increase the expected risk of exposure to the investigational vaccine, compromise the safety of the participant, or interfere with any aspect of study conduct or interpretation of results. This will include asthma and any thrombocytopenia or bleeding disorder contraindicating IM vaccination.
2. Presence of self-reported or medically documented significant medical or psychiatric condition(s).
3. Presence of an acute illness, as determined by the participating site PI or appropriate sub-PI, with or without fever (temperature ≥ 38.0 ºC) within 72 hours prior to each vaccination.
4. Presence of birthmarks, tattoos, wound, or other skin conditions over the deltoid region of both arms that, in the PI's opinion, could reasonably obscure and interfere with evaluation of local ISRs.
5. Inadequate venous access to allow collection of blood samples.
6. Breastfeeding or planning to breastfeed from the time of the first vaccination through 60 days after the last vaccination, or pregnant as confirmed by a positive serum β-HCG pregnancy test at Screening or positive urine pregnancy test at subsequent clinic visits at timepoints as delineated in the schedule of assessments.
7. Received any prophylactic or therapeutic vaccine, or licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication, within 4 weeks of first vaccination or 5 half-lives (whichever is longer), or anticipate to do so in the follow-up period defined for this study.
8. Participant has previously participated in an investigational study involving LNPs (a component of the investigational vaccine assessed in this trial).
9. History of severe allergy (requiring hospital care), severe reaction to any drug or prior vaccination, or any known or suspected allergies or sensitivities to any component of the investigational vaccine or placebo.
10. History of ever had an anaphylaxis reaction to food, medication or vaccination.
11. Participant is immunosuppressed as caused by disease (such as HIV).
12. Chronic use (more than 14 continuous days) of or anticipated need to use, within the next 6 months, of any medications that may be associated with impaired immune responsiveness or with immunosuppression.
13. History of hepatitis B or hepatitis C infection.
14. Receipt of immunoglobulins or blood products within 3 months of first vaccination.
15. Requirement for antipyretic or analgesic medication on a daily or every other day basis from enrolment through 72 hours after vaccination.
16. Current use of any prescription or over-the-counter medications within 7 days prior to vaccination, unless approved by the PI.
17. History of alcohol or drug abuse that in the opinion of the PI could affect the participant's safety or compliance with study.
18. Participant unwilling to abstain from blood donation during the course of the study, and/or participation in any research study involving blood sampling (more than 450 mL /unit of blood), or blood donation to any blood bank during the 2 months prior to the Screening visit.
19. Close contact with anyone known to have SARS-CoV-2 infection within 30 days prior to vaccine administration.
20. Positive for SAR-CoV-2 by antibody IgG/IgM and anti spike IgG at screening
21. History of COVID-19 diagnosis (the criteria for COVID-19 diagnosis will follow the local guidelines).
22. On current treatment with investigational agents for prophylaxis of COVID-19.
23. Planning to travel outside Thailand from enrolment through 28 days after the second vaccination.
24. Residing in a nursing home or other skilled nursing facility or having a requirement for skilled nursing care.
25. Is a participant at high risk of SARS-CoV2 exposure in the opinion of the PI (e.g., healthcare workers, active health care workers with direct patient contact, emergency response personnel).

    Elderly Participants (Group 2 of Phase 1) only
26. Chronically smoking (defined as ≥10 Pack years [packs/day × years smoked]) within the 12 months prior to enrolment.
27. Presence of co-morbidities that can be associated with an increased risk of severe COVID-19 Cancer, Chronic kidney diseases, COPD, cardiovascular disease, solid organ transplantation, DM type 2, HT, cerebrovascular disease, Obesity (BMI> 30 kg/m2)

    Participants for Phase 2 only
28. Presence of co-morbidities that can be associated with an increased risk of severe COVID-19 Cancer, Chronic kidney diseases, COPD, cardiovascular disease, solid organ transplantation, DM type 2, uncontrolled HT, cerebrovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Phase 1 and 2: Frequency of Adverse Events | up to Day 50
  Frequency of Adverse Events
Phase 1 and 2: Grade of Adverse Events | up to Day 50
  Grade of Adverse Events
Phase 1 and 2: Frequency of solicited reportable local Adverse Events | during a 7-day follow-up period post each vaccination
  Frequency of solicited reportable local Adverse Events (i.e., pain, tenderness, erythema/redness, induration/swelling, ulceration, scabs, ecchymosis, oedema, itching, paraesthesia, and hypersensitivity)
Phase 1 and 2: Grade of solicited reportable local Adverse Events | during a 7-day follow-up period post each vaccination
  Grade of solicited reportable local Adverse Events: (i.e., pain, tenderness, erythema/redness, induration/swelling, ulceration, scabs, ecchymosis, oedema, itching, paraesthesia, and hypersensitivity)
Phase 1 and 2: Frequency of solicited reportable systemic reactogenicity Adverse Events | during a 7-day follow-up period post each vaccination
  Frequency of solicited reportable systemic Adverse Events: (i.e., headache, fatigue, myalgia, malaise, fever, rigors, arthralgia, nausea/vomiting, diarrhea, light headedness, dizziness, or any other symptoms)
Phase 1 and 2: Grade of of solicited reportable systemic Adverse Events | during a 7-day follow-up period post each vaccination
  Grade of solicited reportable systemic Adverse Events: (i.e., headache, fatigue, myalgia, malaise, fever, rigors, arthralgia, nausea/vomiting, diarrhea, light headedness, dizziness, or any other symptoms)
Phase 1 and 2: Frequency of Serious Adverse Events | up to Day 387
  Frequency of Serious Adverse Events
Phase 1 and 2: Frequency of Medically-Attended Adverse Events | up to Day 387
  Frequency of Medically-Attended Adverse Events
Phase 1 and 2: Frequency of New-Onset Chronic Medical Conditions | up to Day 387
  Frequency of New-Onset Chronic Medical Conditions
Phase 1 and 2: Changes in vital signs | up to Day 50
  Changes in vital signs: (i.e., body temperature, respiratory rate, pulse rate, systolic blood pressure (SBP), and diastolic blood pressure (DBP))
Phase 1 and 2: Changes in physical examinations | up to Day 50
  Changes in physical examinations: (i.e., head, ears, nose, throat, lungs, lymph nodes, heart, abdomen and skin)
Phase 1 and 2: Changes in laboratory measurements | up to Day 50
  Changes in laboratory measurements: (i.e., haemoglobin (Hb), haematocrit (HCT), white blood cells (WBC), neutrophil, lymphocytes, eosinophil, basophil, monocytes, platelet, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, total protein, albumin, lipase, phosphorus, gamma-glutamyl transferase (GGT), glucose, creatinine phosphokinase (CPK), calcium, uric acid, C-reactive protein (CRP), alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), total bilirubin, estimated glomerular filtration rate (eGFR), prothrombin time (PR), partial thromboplastin time (PTT) and international normalized ratio (INR))
Phase 1 and 2: Presence of injection site reactions | up to Day 50
  Presence of injection site reactions
Phase 2: Geometric mean titers (GMT) in SARS-CoV-2-specific serum neutralising antibody levels | at Day 29 (7 days after the second dose)
  Geometric mean titers (GMT) in SARS-CoV-2-specific serum neutralising antibody levels

SECONDARY OUTCOMES:
Phase 1: Geometric mean titers (GMT) in SARS-CoV-2-specific serum neutralising antibody levels | at Day 29 (7 days after the second dose)
  Geometric mean titers (GMT) in SARS-CoV-2-specific serum neutralising antibody levels
Phase 1 and Phase 2: Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2-specific serum neutralising antibody levels | At Day 29
  Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2-specific serum neutralising antibody levels
Phase 1 and Phase 2: Geometric mean fold rises (GMFR) in SARS-CoV-2-specific serum neutralising titers | from baseline to Day 29
  Geometric mean fold rises (GMFR) in SARS-CoV-2-specific serum neutralising titers
Phase 1 and Phase 2: Geometric mean titers (GMT) in SARS-CoV-2 surrogate viral neutralising antibody levels | at Day 29
  Geometric mean titers (GMT) in SARS-CoV-2 surrogate viral neutralising antibody levels
Phase 1 and Phase 2: Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2 surrogate viral neutralising antibody levels | at Day 29
  Proportion of participants who achieved a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2 surrogate viral neutralising antibody levels
Phase 1 and Phase 2: Geometric mean fold rises (GMFR) in SARS-CoV-2 surrogate viral neutralising antibody titers | from baseline to Day 29
  Geometric mean fold rises (GMFR) in SARS-CoV-2 surrogate viral neutralising antibody titers
Phase 1 and Phase 2: Geometric mean titers (GMT) of SARS-Cov2-spike protein-binding IgG antibody | at Day 29
  Geometric mean titers (GMT) of SARS-Cov2-spike protein-binding IgG antibody
Phase 1 and Phase 2: Proportion of participants who seroconverted: achieving a greater than or equal to 4-fold rise in SARS-Cov2-spike protein-binding IgG antibody | from baseline to Day 29
  Proportion of participants who seroconverted: achieving a greater than or equal to 4-fold rise in SARS-Cov2-spike protein-binding IgG antibody
Phase 1 and Phase 2: Geometric mean fold rises (GMFR) in SARS-Cov2-spike protein-binding IgG antibody | from baseline to Day 29
  Geometric mean fold rises (GMFR) in SARS-Cov2-spike protein-binding IgG antibody
Phase 1 and Phase 2: Percentage of participants who have positive specific CD4 T-cell IFNγ ELISpot responses | Day 29
  Percentage of participants who have positive specific CD4 T-cell IFNγ ELISpot responses
Phase 1 and Phase 2: Percentage of participants who have positive specific CD8 T-cell IFNγ ELISpot responses | Day 29
  Percentage of participants who have positive specific CD8 T-cell IFNγ ELISpot responses
Phase 1 and Phase 2: Median number of spot-forming cells (SFC) per 1 million PBMCs | Day 29
  Median number of spot-forming cells (SFC) per 1 million PBMCs
Phase 1 and Phase 2: Percentage of participants who shows positive specific Th1 responses | Day 29
  Percentage of participants who shows positive specific Th1 responses
Phase 1 and Phase 2: Percentage of participants who shows positive specific Th2 responses | Day 29
  Percentage of participants who shows positive specific Th2 responses
Phase 1 and Phase 2: Median percentage specific Th1 responses | Day 29
  Median percentage specific Th1 responses
Phase 1 and Phase 2: Median percentage specific Th2 responses | Day 29
  Median percentage specific Th2 responses

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Study Director — Center of Excellence in Vaccine Research and Development, Faculty of Medicine, Chulalongkorn University
Locations (2):
- Thailand (2):
  - Chula Vaccine Research Center (ChulaCRC) Faculty of Medicine Chulalongkorn University, Bangkok
  - Center of Excellence for Vaccine Trial (Vaccine Trial Centre), Faculty of Tropical Medicine Mahidol University, Bangkok

REFERENCES:
- [Derived] Puthanakit T, Prompetchara E, Gatechompol S, Ketloy C, Thitithanyanont A, Jongkaewwattana A, Buranapraditkun S, Ubolyam S, Kerr SJ, Sophonphan J, Apornpong T, Kittanamongkolchai W, Siwamogsatham S, Sriplienchan S, Patarakul K, Theerawit T, Promsena P, Nantanee R, Manomaisantiphap S, Chokyakorn S, Hong L, Samija M, Montefiori DC, Gao H, Eaton A, Wijagkanalan W, Alameh MG, Weissman D, Ruxrungtham K; ChulaVac001-Phase 2 study team. Phase II prefusion non-stabilised Covid-19 mRNA vaccine randomised study. Sci Rep. 2024 Jan 29;14(1):2373. doi: 10.1038/s41598-023-49653-6. PMID 38287068